CLINICAL TRIAL: NCT06061874
Title: Ga68-labeled Fibroblast Activation Protein Inhibitor-46 (Ga68-FAPI-46) PET/CT for Preoperative Assessment of Peritoneal Carcinomatosis
Brief Title: Ga68-FAPI-46 PET/CT for Preoperative Assessment of Peritoneal Carcinomatosis
Acronym: FAPeCa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IJB-NM-FAPeCa1
Record Dates: First submitted 2023-08-31; First posted 2023-09-29 (Actual); Last update posted 2025-03-31 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Peritoneal Carcinomatosis
Keywords: colorectal cancer; ovarian cancer; peritoneal carcinomatosis; fibroblast activation protein inhibitor; positron emission tomography; FAPI-46; PET; FAPI; PET/CT; fibroblast activation protein
MeSH Terms: conditions — Neoplasms; Peritoneal Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAPI PET/CT (Experimental): Patients with known or suspected peritoneal metastases from colorectal and ovarian cancers scheduled for complete cytoreductive surgery undergo FAPI PET/CT before the planned surgery.
  In the target population, patients receiving neoadjuvant chemotherapy undergo FAPI PET/CT both before and after chemotherapy.
  Interventions: Diagnostic Test: FAPI PET/CT

INTERVENTIONS:
Diagnostic Test: FAPI PET/CT — The radiopharmaceutical 68Gallium-FAPI-46 (FAPI) is applied intravenously for molecular imaging of FAP expression with FAPI PET/CT.

SUMMARY:
This is a prospective, phase II, non-randomized clinical imaging trial. Ga68-FAPI-46 is a novel radiotracer used in PET/CT imaging, targeting a protein of the tumor microenvironment called FAP (Fibroblast activation protein).

The aim of the study is to assess the accuracy of Ga68-FAPI-46 PET/CT for preoperative assessment of peritoneal carcinomatosis in colorectal and ovarian cancer.

DETAILED DESCRIPTION:
Fibroblast activation protein (FAP) is a type II transmembrane glycoprotein expressed on the surface of cancer-associated fibroblasts (CAFs) in the stroma of various tumor entities. Recently, radiolabeled molecules targeting the FAP, called FAP inhibitors (FAPI) labelled with Gallium-68, have been developed for molecular imaging with PET/CT (positron emission tomography/computed tomography). This radiotracer often presents a higher cancer lesion detectability than F18-FDG (fluorodeoxyglucose), partly thanks to its higher tumour-to-background ratio achieved by a low background activity, particularly in the brain, abdominal cavity and liver. These advantages have resulted in a superior sensitivity of Ga68-FAPI PET/CT over F18-FDG and higher SUV (standardized uptake value) in evaluating various types of cancer. In this context, Ga68-FAPI PET/CT seems promising to further study as a clinical imaging modality for preoperative assessment of peritoneal carcinomatosis.

In this study, the investigators correlate Ga68-FAPI PET/CT findings in terms of peritoneal involvement with intraoperative findings based on histopathology and try to find out how accurate Ga68-FAPI PET/CT is for the preoperative assessment of peritoneal carcinomatosis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal and ovarian cancer.
* Known or suspected peritoneal metastases from the tumour of origin.
* Scheduled for peritoneal complete cytoreductive surgery with curative intent with or without neoadjuvant chemotherapy.
* ECOG (Eastern Cooperative Oncology Group) Performance status ≤2.
* Signed written informed consent obtained before any study-specific screening procedures.

Exclusion Criteria:

* Non-resectable extra-abdominal metastasis and/or >3 hepatic metastases on standard work-up
* Known chronic inflammatory conditions including the intestinal system (eg. inflammatory bowel disease, Crohn's disease)
* Pregnant and lactating women
* Previous or concurrent malignancy diagnosed within the last 3 years except adequately treated in situ carcinoma of the cervix uteri and basal or squamous cell skin cancer.
* Subjects with another significant medical condition which, in the investigator's opinion, may interfere with the completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of the Ga68-FAPI PET/CT derived PCI (peritoneal cancer index) score with the intraoperative PCI based on histopathology of resected specimen (the reference standard) | Through completion of post-surgical pathological examination, up to 2 years since the study initiation
  Intraoperative PCI validated by histopathology performed on resected peritoneal metastases obtained during peritoneal cytoreductive surgery/explorative laparoscopy or laparotomy will be correlated with Ga68-FAPI PET/CT derived PCI.

SECONDARY OUTCOMES:
Comparison of PCI obtained with Ga68-FAPI PET/CT to the PCI calculated on standard preoperative imaging. | Through completion of imaging examinations, up to 2 years since the study initiation
  PCI calculated on standard preoperative imaging (MRI and FDG PET/CT) will be correlated with Ga68-FAPI PET/CT derived PCI.
Assessment of the impact of neoadjuvant chemotherapy on the FAPI expression of target lesions at baseline. | Through completion of post-neoadjuvant chemotherapy FAPI PET examination,up to 2 years since the study initiation
  Subgroup: Patients receiving neoadjuvant chemotherapy Treatment-induced change in the total peritoneal tumor volume and uptake intensity of FAPI on PET/CT will be assessed and correlated to histopathological findings.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Flamen, Principal Investigator — Jules Bordet Institute
Locations (1):
- Institut Jules Bordet, Brussels, Belgium